CLINICAL TRIAL: NCT02561702
Title: Mexiletine for Muscle Cramps in Charcot Marie Tooth Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, David Herrmann, Professor, University of Rochester
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RSRB00057653
Record Dates: First submitted 2015-09-24; First posted 2015-09-28 (Estimated); Results first posted 2018-03-26 (Actual); Last update posted 2018-03-26 (Actual); Status verified 2018-02

CONDITIONS: Charcot Marie Tooth Disease
MeSH Terms: conditions — Charcot-Marie-Tooth Disease | interventions — Mexiletine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mexiletine first/placebo second (Experimental): Participants will receive 150 mg of mexiletine by mouth 3 times daily for 5-7 days followed by 7 day washout period and 5-7 days of placebo (240 mg of lactose powder) taken by mouth 3 times daily
  Interventions: Other: Placebo; Drug: Mexiletine
- placebo first/mexiletine second (Experimental): Participants will receive placebo (240 mg of lactose powder) taken by mouth 3 times daily for 5-7 days followed by 7 day washout period and 5-7 days of 150 mg of mexiletine by mouth 3 times daily
  Interventions: Other: Placebo; Drug: Mexiletine

INTERVENTIONS:
Other: Placebo — 240 mg lactose powder in a size 3 capsule taken by mouth 3 times daily for 5-7 days
  Other Names: lactose powder
Drug: Mexiletine — 150 mg Mexiletine taken by mouth in capsule form 3 times daily for 5-7 days

SUMMARY:
Charcot Marie Tooth Disease is a family of inherited peripheral neuropathies, with over 70 causative genes identified to date.1-4 Muscle cramps are frequent in CMT, affecting up to 85% of patients with some subtypes of CMT. These cramps impact quality of life and have been identified as an important therapeutic target for clinical trials in CMT.1-4 There is no FDA approved treatment for muscle cramps.5 Mexiletine is a sodium channel blocker approved for treatment of arrhythmias. As a sodium channel blocker, mexiletine offers the promise of effective therapy for muscle cramps.

DETAILED DESCRIPTION:
This study will provide data on the short term efficacy of oral mexiletine in helping to prevent muscle cramps in adults with CMT. The study will also assess the short-term safety and tolerability of low dose mexiletine in adults with CMT.

ELIGIBILITY:
Inclusion Criteria:

* The subject has known CMT, previously diagnosed by a neurologist with subspeciality expertise in neuromuscular disorders/peripheral neuropathy. The diagnosis of CMT relies on a combination of clinical history (including family history), neurological examination electrophysiological features, and prior genetic testing results.

  * The subject is at least 18 years old, and has signed the Informed Consent Form.
  * The subject is ambulatory (cane, walker, orthoses allowed).
  * The subject has experienced muscle cramps and has known provokable hamstring or calf muscle cramps on MVC.
  * The subject has a reliable method of birth control (if a female subject of child bearing potential). Reliable birth control is defined as Hormonal contraception Intrauterine contraception/device Any two barrier methods (combination of male or female condom with diaphragm sponge or cervical cap) together with spermicidal foam/gel/film/cream/suppository True abstinence

Exclusion Criteria:

* The subject has a known neuropathy from another source (e.g., diabetes, drug induced, alcohol, etc.).

  * The subject has an untreated medical disorder known to predispose to muscle cramps
  * The subject is pregnant or nursing, has a known mexiletine allergy or has taken mexiletine in the past 12 weeks.
  * The subject is participating in another therapeutic trial.
  * The subject has second or 3rd degree heart block, atrial flutter/fibrillation, ventricular arrhythmias, or is receiving treatment of a cardiac arrhythmia.
  * The subject is currently taking another agent for muscle cramps or a muscle relaxant (e.g., benzodiazepine, baclofen, tizanidine, soma, meprobromate).
  * The subject is on another sodium channel blocker or medication that precludes administration of mexiletine.
  * The subject has known diabetes mellitus, liver or kidney disease requiring ongoing treatment, untreated thyroid dysfunction, symptomatic cardiomyopathy, or symptomatic coronary artery disease.
  * The subject, in the opinion of the investigator, is unsuitable for enrollment for any other reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-09; Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Herrmann, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: First Intervention
Arm/Group | Mexiletine First/Placebo Second | Placebo First/Mexiletine Second
Started | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0
Period: Washout
Arm/Group | Mexiletine First/Placebo Second | Placebo First/Mexiletine Second
Started | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Mexiletine First/Placebo Second | Placebo First/Mexiletine Second
Started | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Decrease in Cramp Duration
Description: Participant will be evaluated for muscle cramps 120 minutes following a single dose of oral mexiletine. The Clinical Evaluator applied pressure to provoke hamstring cramps bilaterally, one at a time 2 hours after dose. The cramp duration in seconds of the right hamstring was used.
Time Frame: 120 minutes
Measure: Number; unit: participants
Groups:
- Mexiletine: Participants will receive 150 mg of mexiletine by mouth 3 times daily for 5-7 days followed by 7 day washout period and 5-7 days of placebo (240 mg of lactose powder) taken by mouth 3 times daily
  Placebo: 240 mg lactose powder in a size 3 capsule taken by mouth 3 times daily for 5-7 days
  Mexiletine: 150 mg Mexiletine taken by mouth in capsule form 3 times daily for 5-7 days
- Placebo: Participants will receive placebo (240 mg of lactose powder) taken by mouth 3 times daily for 5-7 days followed by 7 day washout period and 5-7 days of 150 mg of mexiletine by mouth 3 times daily
  Placebo: 240 mg lactose powder in a size 3 capsule taken by mouth 3 times daily for 5-7 days
  Mexiletine: 150 mg Mexiletine taken by mouth in capsule form 3 times daily for 5-7 days
Arm/Group | Mexiletine | Placebo
Number analyzed (Participants) | 4 | 4
participants | 2 | 0

2. Primary Outcome: Number of Participants With a Decrease in Cramp Intensity
Description: Participant will be evaluated for muscle cramps 120 minutes following a single dose of oral mexiletine. The Clinical Evaluator applied pressure to provoke hamstring cramps bilaterally, one at a time 2 hours after dose. The cramp intensity of the right hamstring was reported by the subject on a scale of 1-10 with 1 being weak and 10 being severe.
Time Frame: 120 minutes
Measure: Number; unit: participants
Arm/Group | Mexiletine | Placebo
Number analyzed (Participants) | 4 | 4
participants | 1 | 2

ADVERSE EVENTS:
Arm/Group | Mexiletine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes